CLINICAL TRIAL: NCT04998955
Title: Maximal Strength Training in Patients With Inflammatory Rheumatic Disease: Implications for Physical Function and Quality of Life
Brief Title: MST in Patients With Inflammatory Rheumatic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molde University College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HHRevma2 - MST
Record Dates: First submitted 2021-07-12; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Inflammatory Rheumatism
Keywords: Maximal strength; Quality of life; Heavy resistance training; Rate of force development; Rehabilitation
MeSH Terms: conditions — Rheumatic Fever

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was blinded with regards to which intervention group the participants had been assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MST group (Experimental): Exercise intervention, 20 supervised MST sessions
  Interventions: Behavioral: Maximal strength training
- Control group (No Intervention): IRD patient controls

INTERVENTIONS:
Behavioral: Maximal strength training — Exercise intervention utilizing 4 x 4 repetitions heavy resistance training
  Arms: MST group

SUMMARY:
The purpose of this study is to investigate the feasibility of 10 weeks of maximal strength training (MST) in patients with inflammatory rheumatic disease. As well as the effects of MST on maximal strength, rate of force developement and quality of life in this patient population.

DETAILED DESCRIPTION:
Patients with inflammatory rheumatic diseases (IRD) such as rheumatoid arthritis, spondyloarthritis and systemic lupus erythematosus have reduced strength and muscle mass in the lower extremities compared to healthy control groups. This attenuation results in impaired physical function and health-related quality-of-life. Maximum muscle strength is an important indicator of total mortality, even when adjusted for cardiovascular health. Therefore, international guidelines encourage strength training since it has been demonstrated that resistance exercise using moderate loads (≤80% of one repetition maximum; 1RM) result in improved strength and function without worsening pain or disease activity.

In this trial patients are randomized into either a maximal strength training (MST) intervention group or a control group. The intervention period will last 10 weeks. The MST group will perform two supervised MST sessions per week, on non-consecutive days, in a seated horizontal leg press apparatus. The control group will continue with their existing activity routines. One MST session consist of 4 series of 4 repetitions maximum (4RM) utilizing heavy loads (~90 % of 1RM), separated by 3 minutes break and lasts approximately 15-20 minutes. The MST intervention follows the principle of linear progression continuously adjusting the resistance to achieve the targeted 4RM training load. The control group will be given supervised introduction to effective strength training after the intervention period.

The purpose of this intervention is to evaluate the feasibility of the highly potent MST intervention and its impact on 1RM, rate of force development (RFD) and quality of life in the IRD patient population. MST has been documented to yield almost twice the increase in both 1RM and RFD as conventional strength training performed with moderate resistance. However, it is uncertain if MST is well tolerated by the IRD patient population which is characterized by having pain, stiffness, and joint swelling. Before and after the training period, identical testing (approximately 60 min) will be performed by both intervention groups. The testing will include measurements of maximal oxygen uptake in an endurance test as well as maximal muscle strength, recorded as 1RM, and dynamic RFD both carried out in a horizontal leg press apparatus. Additionally, quality of life questionnaires will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory rheumatic disease

Exclusion Criteria:

* Inability to complete the testing procedures
* Pregnancy
* Not able to perform exercise intervention
* Planed surgeries or other plans during initial exercise intervention period than directly will effect the testing or training.
* unstable ischemic heart disease
* unstable aortic stenosis or aneurysm
* Less than 80% compliance of planned training sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Change in physiological measure assesed in the horizontal leg press apparatus | At baseline and after 10 weeks.
  Maximal strength; one repetition maximum (measured in kg)

SECONDARY OUTCOMES:
Change in health-related quality of life assessed by Norwegian RAND-36 | At baseline and after 10 weeks
  Questionnaire scoring on a 0-100 scale with higher scores identifying better outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Jan Helgerud, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Myworkout - Medical Rehabilitation Clinic, Trondheim, Please Select, Norway

REFERENCES:
- [Derived] Haglo H, Berg OK, Hoff J, Helgerud J, Wang E. Maximal strength training in patients with inflammatory rheumatic disease: implications for physical function and quality of life. Eur J Appl Physiol. 2022 Jul;122(7):1671-1681. doi: 10.1007/s00421-022-04948-w. Epub 2022 Apr 19. PMID 35438424